CLINICAL TRIAL: NCT00003361
Title: Phase II Study With Decitabine (5-aza-2'-Deoxycytidine, DAC) in Myelodysplastic Syndromes
Brief Title: Decitabine in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-98017; CDR0000066343 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1444
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of decitabine in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response of patients with myelodysplastic syndromes (including chronic myelomonocytic leukemia) to decitabine.

OUTLINE: This is an open label, multicenter study. Patients are stratified by disease (low risk myelodysplastic syndrome (MDS) vs. high risk MDS vs. chronic myelomonocytic leukemia). Patients receive decitabine as a 4 hour infusion every 8 hours on days 1-3. Treatment continues every 6-8 weeks for 4-6 courses. Patients are followed at 6 and 12 months.

PROJECTED ACCRUAL: Approximately 75 patients will be accrued for this study over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven myelodysplastic syndrome Refractory anemia (RA) RA with ringed sideroblasts (RARS) RA with excess blasts (RAEB) RAEB in transformation Chronic myelomonocytic leukemia (CMML) RA and RARS: Platelet count less than 50,000/mm3 CMML: If WBC greater than 10,000/mm3, then must have at least 8% monocytes in the blood or marrow

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease Other: No active or uncontrolled infection Not pregnant or nursing Fertile patients must use effective contraception No other active cancer except skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than one prior chemotherapy regimen for myelodysplastic syndromes At least 3 weeks since chemotherapy and recovered No prior high-dose cytarabine (at least 0.5 g/m2 for at least 4 doses) Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1998-04; Primary Completion 2003-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Nimer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas